CLINICAL TRIAL: NCT04352803
Title: IV Infusion of Autologous Adipose Derived Mesenchymal Cells for Abatement of Respiratory Compromise in SARS-CoV-2 Pandemic (COVID-19)
Brief Title: Adipose Mesenchymal Cells for Abatement of SARS-CoV-2 Respiratory Compromise in COVID-19 Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneris Medical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COVID-MSCIV
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Covid-19 Pneumonia; Cyotokine Storm
Keywords: Coronavirus; SARS-CoV-2; ARDS; Pandemic
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: This is an Interventional, Prospective, Open label (Voluntary Assignment), single to multiple center expansion, unmatched controlled, Sequentially Interim analysis tested Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Adipose Derived Mesenchymal Cells (Experimental): Conventional treatment plus MSC's IV
  Interventions: Biological: Autologous Adipose MSC's
- Untreated (No Intervention): Conventional treatment only

INTERVENTIONS:
Biological: Autologous Adipose MSC's — Autologous Adipose Derived Mesenchymal Cells 500,000/kg IV
  Arms: Autologous Adipose Derived Mesenchymal Cells

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of autologous adipose-derived mesenchymal cells for treating confirmed or suspected patients with SARS-CoV-2 and compromised respiratory function requiring hospitalization.

The hypothesis of the Study is autologous adipose-derived mesenchymal cells given IV to eligible patients will improve clinical outcomes of COVID 19 positive patients with severe pneumonia or ARDS by reducing or avoiding cytokine storm.

DETAILED DESCRIPTION:
While most patients with SARS-CoV-2 present with mild respiratory disease with the most common symptoms of fever and cough, approximately 14 % progress to severe pneumonia and ARDS.

The overall mortality rate is 2% but varies by country and age of the patient.

In COVID-19 ARDS standard supportive care and treatment for underlying illnesses remain the mainstay with limited success.

Numerous antiviral medications including remdesivir, lopinavir-ritonavir or lopinavir-ritonavir and interferon Beta-1a are in clinical trials but safety and efficacy remain unclear.

Inflammation associated with a cytokine storm begins at a local site and spreads throughout the body via systemic circulation. The lungs and other organs are damaged with progressive inflammation.

Mesenchymal cells offer the potential to treat viral infection both directly and through reducing the immune response. MSCs play a role as an immunomodulator, which is safe and effective as demonstrated in numerous clinical trials.

Mesenchymal cells are a potential privileged cell-based therapy in SARS-CoV-2. MSCs derived extracellular vesicles have demonstrated comparable and sometimes more effective effects in ameliorating lung inflammation and injury.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of and less than 90
2. COVID 19 diagnosis confirmed
3. Ability to give informed consent
4. Hospitalized

Exclusion Criteria:

1. Mild Illness

   1. Patients with uncomplicated upper respiratory tract viral infection, may have non-specific symptoms such as fever, fatigue, cough (with or without sputum production), anorexia, malaise, muscle pain, sore throat, dyspnea, nasal congestion, or headache. Rarely, patients may also present with diarrhea, nausea and vomiting.
   2. The elderly and immunosuppressed candidates may present with atypical symptoms. Symptoms due to physiologic adaptations of pregnancy or adverse pregnancy events, such as e.g. dyspnea, fever, GI-symptoms or fatigue, may overlap with COVID-19 symptoms. Still, they will be excluded, unless they progress to Inclusion Criteria within 72 hours from recruitment.
2. Pneumonia (uncomplicated):

   a. Adults with pneumonia but no signs of severe pneumonia AND NO need for supplemental oxygen
3. Reported pregnant or positive pregnancy test
4. Other chronic respiratory disorders such as COPD, emphysema, lung cancer, or cystic fibrosis
5. BMI lower than 21
6. Skinfold test < 3 cm at harvest area
7. Patients with Do-Not-Resuscitate orders that limit mechanical ventilation assistance in place at hospital admission
8. Males and females < 18 years of age
9. Patients who are currently breastfeeding
10. Co-Infection of HIV, tuberculosis, influenza virus, adenovirus and other respiratory infection viruses.
11. History of systemic malignant neoplasms within the last 5 years.
12. Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason
13. Participating in another clinical research study
14. History of Bleeding disorder which in PI's opinion would render the patient unsuitable for the study
15. PT (plasma) < 9 or >11.6 seconds and in the opinion of the PI and attending physician that lipoaspiration would be contraindicated. May be eligible for re-screening if coagulopathy improves within 72 hours of consent
16. PTT < 23 or >32 seconds and in the opinion of the PI and attending physician that lipoaspiration would be contraindicated. May be eligible for re-screening if coagulopathy improves within 72 hours of consent
17. Platelets count less than 70,0000
18. History of DVT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Safety - Incidence of unexpected adverse events | up to 28 days
  Incidence of unexpected adverse events within 28 days following IV administration of MSCs.
Efficacy - Frequency of progression to mechanical ventilation | up to 28 days
  Changes in progression or rate of subjects progressing to mechanical ventilation
Efficacy - Changes in length of mechanical ventilation | up to 28 days
  Changes in time subjects remain on mechanical ventilation
Efficacy - Changes in length of weaning of mechanical ventilation | up to 28 days
  Changes in length of time subjects wean off of mechanical ventilation
Efficacy - Changes in length of hospital stay | up to 28 days
  Length of Hospital Stay
Efficacy - Changes in mortality rate | up to 28 days
  Mortality rate from all causes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Mar;55(3):105924. doi: 10.1016/j.ijantimicag.2020.105924. Epub 2020 Feb 17. PMID 32081636
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Leng Z, Zhu R, Hou W, Feng Y, Yang Y, Han Q, Shan G, Meng F, Du D, Wang S, Fan J, Wang W, Deng L, Shi H, Li H, Hu Z, Zhang F, Gao J, Liu H, Li X, Zhao Y, Yin K, He X, Gao Z, Wang Y, Yang B, Jin R, Stambler I, Lim LW, Su H, Moskalev A, Cano A, Chakrabarti S, Min KJ, Ellison-Hughes G, Caruso C, Jin K, Zhao RC. Transplantation of ACE2- Mesenchymal Stem Cells Improves the Outcome of Patients with COVID-19 Pneumonia. Aging Dis. 2020 Mar 9;11(2):216-228. doi: 10.14336/AD.2020.0228. eCollection 2020 Apr. PMID 32257537
- [Background] Mohammadzadeh A, Pourfathollah AA, Shahrokhi S, Hashemi SM, Moradi SL, Soleimani M. Immunomodulatory effects of adipose-derived mesenchymal stem cells on the gene expression of major transcription factors of T cell subsets. Int Immunopharmacol. 2014 Jun;20(2):316-21. doi: 10.1016/j.intimp.2014.03.003. Epub 2014 Apr 3. PMID 24704622
- [Background] Zuk PA, Zhu M, Mizuno H, Huang J, Futrell JW, Katz AJ, Benhaim P, Lorenz HP, Hedrick MH. Multilineage cells from human adipose tissue: implications for cell-based therapies. Tissue Eng. 2001 Apr;7(2):211-28. doi: 10.1089/107632701300062859. PMID 11304456